CLINICAL TRIAL: NCT05966155
Title: A Depression and Opioid Pragmatic Trial in Pharmacogenetics
Brief Title: A Depression and Opioid Pragmatic Trial in Pharmacogenetics (Depression Trial)
Acronym: ADOPT PGx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Human Genome Research Institute (NHGRI) (NIH); University of Florida (Other); Vanderbilt University Medical Center (Other); Indiana University School of Medicine (Other); Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO00104948_C; U01HG010225 (NIH)
Record Dates: First submitted 2023-07-21; First posted 2023-07-28 (Actual); Results first posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Depression
Keywords: Pharmacogenetic; CYP2D6; CYP2C19
MeSH Terms: conditions — Depression | interventions — Pharmacogenomic Testing

STUDY DESIGN:
Intervention Model Description: Immediate vs. delayed pharmacogenetic testing and genotype-guided pain or depression therapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Depression - Immediate PGx Testing (Experimental): Immediate genetic testing of CYP2D6 and CYP2C19 and clinical decisions support for antidepressant prescribing to the healthcare provider
  Interventions: Other: Pharmacogenetic testing; Other: Clinical decisions support
- Depression - Delayed PGx Testing (Other): Delayed genetic testing of CYP2D6 and CYP2C19 and return of results after the conclusion of the 6-month follow-up period
  Interventions: Other: Pharmacogenetic testing

INTERVENTIONS:
Other: Pharmacogenetic testing — Genetic testing of CYP2D6 and CYP2C19
Other: Clinical decisions support — Prescribing recommendations to the provider based on the pharmacogenetic testing results
  Arms: Depression - Immediate PGx Testing

SUMMARY:
This study is comprised of three separate pharmacogenetic trials grouped into a single protocol due to similarities in the intervention, the hypotheses, and the trial design. The three trials are the Acute Pain Trial, the Chronic Pain Trial, and the Depression Trial. Participants can enroll in only one of the three trials. All three trials were registered on ClinicalTrials.gov under NCT04445792. In July 2023 each of the three treatment trials was registered under a separate NCT# and NCT04445792 was converted to a screening record per recent guidance on master protocol research programs (MPRPs). This record is specific to the Depression Trial within the ADOPT-PGx protocol.

The Depression Trial is a prospective, multicenter, two arm randomized pragmatic trial. Participants meeting eligibility criteria will be randomly assigned to either immediate pharmacogenetic testing and genotype-guided anti-depressant therapy (Intervention arm) or standard care with 6-month delayed pharmacogenetic testing (Control arm). The investigators will test the hypothesis that pharmacogenetic testing and genotype-guided anti-depressant therapy will reduce depression symptoms in participants who's body processes some anti-depressants faster or slower than normal.

DETAILED DESCRIPTION:
Pain and depression are conditions that impact substantial proportions of the US population. Finding safe and effective drug therapies for both conditions is challenging. In the case of treatment for acute and chronic pain, the challenge is finding effective therapy while minimizing adverse effects or opioid addiction (and the ensuing consequences). For depression, there are few clinically relevant predictors of successful treatment leading to multiple trials of inadequate therapy for some patients. Both opioid and antidepressant prescriptions can be guided by pharmacogenetics (PGx) data based on existing guidelines from the Clinical Pharmacogenetics Implementation Consortium (CPIC).

This study is designed to evaluate the impact of pharmacogenetic testing and genotype-guided pain or anti-depressant therapy on pain control or depression symptoms in a pragmatic setting.

The rationale for examining a genotype-guided approach to acute and chronic pain management is based on the importance of CYP2D6 for the bioactivation of tramadol, codeine, and hydrocodone and data from a pilot study supporting improved pain control in intermediate and poor CYP2D6 metabolizers in the genotype-guided arm who are taking these drugs at baseline. Similarly, the rationale for examining a genotype-guided approach to depression medication therapy is based on the demonstrated role of CYP2D6 in the bio inactivation and CYP2C19 oxidation of select, commonly used SSRIs. Secondly, data from industry sponsored trials support the hypothesis of improved depression symptom control in a genotype-guided arm.

Study objectives:

Determine if genotype-guided dosing or selection of antidepressants among participants with at least 3 months of depressive symptoms who require new or revised antidepressant therapy leads to improved control of depression, compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

Depression Trial

* Age ≥ 8 years
* English speaking or Spanish speaking
* Patients followed at psychiatry clinics or primary care clinics at an enrolling site (such as, but not limited to, Internal Medicine, Family Medicine, or Pediatrics)
* Documentation of depression and/or provider report of depression
* Evidence of depressive symptoms for at least 3 months based on patient interview or documentation in electronic health records
* Recent initiation of SSRI therapy, recent revised SSRI therapy, or anticipated need for revised or new SSRI therapy per health care provider

Exclusion Criteria

Trial-wide:

* Life expectancy less than 12 months
* Are too cognitively impaired to provide informed consent and/or complete study protocol
* Are institutionalized or too ill to participate (i.e. mental or nursing home facility or incarcerated)
* Have a history of allogeneic stem cell transplant or liver transplant
* People with prior clinical pharmacogenetic test results for genes relevant for the study in which they will enroll (CYP2D6 for the pain studies and CYP2D6 or CYP2C19 for depression) or already enrolled in an ADOPT PGx trial

Depression Trial

* Plan to move out of the area within 6 months of enrollment
* Have active psychosis or diagnosed psychotic disorders (schizophrenia, schizoaffective disorder, delusional disorder, psychotic depression, substance induced psychosis, schizophreniform disorder)
* Have dementia or other neurocognitive disorders due to any cause, such as Alzheimer's disease, vascular/subcortical, lewy body disease, frontotemporal lobar degeneration
* Have cognitive developmental delay and/or cognitive disability, including autism spectrum disorders (Note: ADHD is not an exclusion criteria)
* Has a seizure disorder
* Have bipolar disorder

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1572 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2024-04-27 (Actual); Study Completion 2024-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hrishikesh Chakraborty, Study Director — Duke University; Josh F. Peterson, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (14):
- United States (14):
  - Nemours Children's Health System, Wilmington, Delaware
  - University of Florida - Gainesville, Gainesville, Florida
  - Nemours Children's Health System, Jacksonville, Florida
  - University of Florida - Jacksonville, Jacksonville, Florida
  - Nemours Children's Health System, Orlando, Florida
  - Eskenazi Health, Indianapolis, Indiana
  - Indiana University, Indianapolis, Indiana
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - The Institute for Family Health, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Sanford Health, Fargo, North Dakota
  - Meharry Medical College, Nashville, Tennessee
  - Nashville General Hospital, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hines LJ, Wilke RA, Myers R, Mathews CA, Liu M, Baye JF, Petry N, Cicali EJ, Duong BQ, Elwood E, Hulvershorn L, Nguyen K, Ramos M, Sadeghpour A, Wu RR, Williamson L, Wiisanen K, Voora D, Singh R, Blake KV, Murrough JW, Volpi S, Ginsburg GS, Horowitz CR, Orlando L, Chakraborty H, Dexter P, Johnson JA, Skaar TC, Cavallari LH, Van Driest SL, Peterson JF; IGNITE Pragmatic Trials Network. Rationale and design for a pragmatic randomized trial to assess gene-based prescribing for SSRIs in the treatment of depression. Clin Transl Sci. 2024 Jun;17(6):e13822. doi: 10.1111/cts.13822. PMID 38860639
- See also: Rationale and design for a pragmatic randomized trial to assess gene-based prescribing for SSRIs in the treatment of depression — http://pubmed.ncbi.nlm.nih.gov/38860639/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This record is specific to the Depression Trial within the ADOPT PGx protocol. It only contains the participants consented to the Depression Trial.
Pre-assignment Details: There were 1572 participants consented into the Depression trial. 112 consented participants were not randomized into the trial and were not assigned to a treatment arm. The 1460 randomized participants will be described moving forward.
Period: Overall Study
Arm/Group | Depression - Immediate PGx Testing | Depression - Delayed PGx Testing
Started | 727 | 733
Completed | 654 | 653
Not Completed | 73 | 80
Not completed — Death | 1 | 2
Not completed — Lost to Follow-up | 63 | 67
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 8 | 9
Not completed — Enrolled Erroneously | 0 | 1
Not completed — Follow-up Incorrectly Scheduled | 0 | 1

BASELINE CHARACTERISTICS:
Population: ITT refers to the Intent To Treat population, while mITT, a subset of ITT, refers to the modified Intent To Treat population. The mITT population is the primary analytical population for the Depression Trial and includes participants who have a CYP2D6 PM, UM or NM-UM phenotype or a CYP2C19 PM, RM, or UM phenotype.
Groups:
- Total: Total of all reporting groups
Arm/Group | Depression - Immediate PGx Testing | Depression - Delayed PGx Testing | Total
Number analyzed (Participants) | 727 | 733 | 1460
Age, Categorical [Count of Participants; unit: Participants] — Population: Intent to Treat Population
  Participants
    <=18 years | 110 | 111 | 221
    Between 18 and 65 years | 550 | 539 | 1089
    >=65 years | 67 | 83 | 150
Age, Categorical [Count of Participants; unit: Participants] — Population: Modified Intent to Treat Population
  Participants
    number analyzed (Participants) | 351 | 341 | 692
    <=18 years | 49 | 48 | 97
    Between 18 and 65 years | 273 | 255 | 528
    >=65 years | 29 | 38 | 67
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Intent to Treat Population
  Participants
    Female | 552 | 544 | 1096
    Male | 175 | 189 | 364
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Modified Intent to Treat Population
  Participants
    number analyzed (Participants) | 351 | 341 | 692
    Female | 266 | 248 | 514
    Male | 85 | 93 | 178
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Intent to Treat Population
  Participants
    Hispanic or Latino | 95 | 96 | 191
    Not Hispanic or Latino | 621 | 629 | 1250
    Unknown or Not Reported | 11 | 8 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Modified Intent to Treat Population
  Participants
    number analyzed (Participants) | 351 | 341 | 692
    Hispanic or Latino | 38 | 54 | 92
    Not Hispanic or Latino | 311 | 285 | 596
    Unknown or Not Reported | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Intent to Treat Population
  Participants
    American Indian or Alaska Native | 4 | 3 | 7
    Asian | 17 | 23 | 40
    Native Hawaiian or Other Pacific Islander | 3 | 3 | 6
    Black or African American | 121 | 110 | 231
    White | 465 | 493 | 958
    More than one race | 27 | 30 | 57
    Unknown or Not Reported | 90 | 71 | 161
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Modified Intent to Treat Population
  Participants
    number analyzed (Participants) | 351 | 341 | 692
    American Indian or Alaska Native | 2 | 2 | 4
    Asian | 5 | 10 | 15
    Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
    Black or African American | 60 | 52 | 112
    White | 235 | 228 | 463
    More than one race | 16 | 15 | 31
    Unknown or Not Reported | 32 | 34 | 66
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 727 | 733 | 1460

OUTCOME MEASURES:

1. Primary Outcome: Change in Depression Symptom Control as Measured by PROMIS (Patient-Reported Outcomes Measurement Information System)
Description: The 8-item PROMIS Emotional Distress Depression 8b and PROMIS Pediatric Depression Symptoms 8a questionnaire assess the extent to which participants experience depression symptoms over the past 7 days using a 5-point Likert scale. The responses to the 8 questions are converted to T-scores using the health measures assessment center scoring service. Pediatric T-scores are cross walked to adult T-scores using the cross walk published in Reeve et al 2016. Cross walked T-scores range from 37.1 to 80.9, higher scores correspond with higher levels of depression symptoms. Changes in T-scores from baseline to 3-months range from -43.8 to 43.8. Negative values of change in T-score correspond to symptom improvement, 0 corresponds to no change in depression T-scores, and positive change in depression T-scores correspond to symptom worsening at 3 months compared to baseline.
Time Frame: Baseline to 3 months
Population: Modified intent to treat (mITT) population consisting of participants with a CYP2C19 poor, rapid, or ultra-rapid metabolizer phenotype or a CYP2D6 poor or ultra-rapid metabolizer phenotype. All mITT participants with completed PROMIS Depression surveys at both baseline and 3 months are included. Participants with missing PROMIS depression surveys at either baseline or 3-months are excluded.
Measure: Mean (Standard Deviation); unit: T-score
Groups:
- Depression - Immediate PGx Testing (Modified Intent to Treat, mITT): Immediate genetic testing of CYP2D6 and CYP2C19 and clinical decisions support for antidepressant prescribing to the healthcare provider
- Depression - Delayed PGx Testing (Modified Intent to Treat, mITT): Delayed genetic testing of CYP2D6 and CYP2C19 and return of results after the conclusion of the 6-month follow-up period
Arm/Group | Depression - Immediate PGx Testing (Modified Intent to Treat, mITT) | Depression - Delayed PGx Testing (Modified Intent to Treat, mITT)
Number analyzed (Participants) | 329 | 320
T-score | -4.3 (8.4) | -4.0 (8.1)
Statistical Analysis 1: Comparison: Depression - Immediate PGx Testing (Modified Intent to Treat, mITT) vs Depression - Delayed PGx Testing (Modified Intent to Treat, mITT); Test type: Superiority; p = 0.677, t-test, 2 sided; Mean Difference (Final Values) = -0.27, 95% CI 2-sided [-1.54 to 1.00]

2. Secondary Outcome: Change in Depression Symptomatology as Measured by Patient Health Questionnaire (PHQ-8)
Description: The 8-item PHQ-8 Questionnaire assesses severity of depression over the past 2 weeks using a 4-point scale indicating frequency of depression symptoms: not at all, several days, more than half the days, or nearly every day. The 8 questions are converted to a score ranging from 0 (not at all for all 8 symptoms) to 24 (nearly every day for all 8 symptoms). Changes in PHQ-8 scores from baseline to 3-months range from -24 to 24 and negative values of change in PHQ-8 correspond to improvement in depression at 3 months compared to baseline.
Time Frame: Baseline to 3 months
Population: Modified ITT population consisting of participants with a CYP2C19 poor, rapid, or ultra-rapid metabolizer phenotype or a CYP2D6 poor or ultra-rapid metabolizer phenotype. All mITT participants with completed PHQ-8 surveys at both baseline and 3 months are included. Participants with missing PHQ-8 surveys at either baseline or 3-months are excluded.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Depression - Immediate PGx Testing (Modified Intent to Treat, mITT) | Depression - Delayed PGx Testing (Modified Intent to Treat, mITT)
Number analyzed (Participants) | 327 | 320
score on a scale | -3.3 (5.2) | -2.7 (4.8)
Statistical Analysis 1: Comparison: Depression - Immediate PGx Testing (Modified Intent to Treat, mITT) vs Depression - Delayed PGx Testing (Modified Intent to Treat, mITT); Test type: Superiority; p = 0.1264, t-test, 2 sided; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-1.4 to 0.2]

3. Secondary Outcome: Side Effect Burden
Description: An 8-item survey was developed to assess the severity of 8 depression medication side effects, using a 4-point scale for rating severity of the side effect: none, mild, moderate, severe. The 8 questions are converted to a side effect burden score ranging from 0 (none for all 8 side effects) to 24 (severe for all 8 side effects). Higher values correspond with more side effects and with higher severity.
Time Frame: 3 months
Population: Modified intent to treat (mITT) population consisting of participants with a CYP2C19 poor, rapid, or ultra-rapid metabolizer phenotype or a CYP2D6 poor or ultra-rapid metabolizer phenotype. All mITT participants with completed medication side effect surveys at 3 months are included. Participants with missing side effect surveys at 3-months are excluded.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Depression - Immediate PGx Testing (Modified Intent to Treat, mITT) | Depression - Delayed PGx Testing (Modified Intent to Treat, mITT)
Number analyzed (Participants) | 285 | 283
score on a scale | 8.2 (4.3) | 7.8 (4.5)
Statistical Analysis 1: Comparison: Depression - Immediate PGx Testing (Modified Intent to Treat, mITT) vs Depression - Delayed PGx Testing (Modified Intent to Treat, mITT); Test type: Superiority; p = 0.3692, t-test, 2 sided; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-0.4 to 1.1] — The by-group means and the estimated mean difference are independently rounded to the nearest tenth. As a result, the mean difference it not exactly equivalent to the difference in the two reported means

4. Secondary Outcome: Medication Non-Adherence as Measured by the Voils Medication Adherence Survey
Description: Medication adherence level, non-adherent / adherent, derived from the Voils Medication Adherence survey. Reported as the number of participants who were non-adherent.
Time Frame: 3 months
Population: Modified intent to treat (mITT) population consisting of participants with a CYP2C19 poor, rapid, or ultra-rapid metabolizer phenotype or a CYP2D6 poor or ultra-rapid metabolizer phenotype. All mITT participants with 2 or more Voils survey questions completed at 3 months are included. Participants with fewer than 2 completed Voils survey questions are excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Depression - Immediate PGx Testing (Modified Intent to Treat, mITT) | Depression - Delayed PGx Testing (Modified Intent to Treat, mITT)
Number analyzed (Participants) | 323 | 317
Participants | 142 | 137
Statistical Analysis 1: Comparison: Depression - Immediate PGx Testing (Modified Intent to Treat, mITT) vs Depression - Delayed PGx Testing (Modified Intent to Treat, mITT); Test type: Superiority; p = 0.8492, Chi-squared

5. Secondary Outcome: Number of Participants With Depression Remission as Measured by PROMIS (Patient-Reported Outcomes Measurement Information System)
Description: Remission is defined as whether or not the summed raw responses to the PROMIS emotional distress depression survey is ≤ 16, corresponding to a participant respond "rarely" or "never" to most or all questions.
Time Frame: 6 months
Population: Modified intent to treat (mITT) population consisting of participants with a CYP2C19 poor, rapid, or ultra-rapid metabolizer phenotype or a CYP2D6 poor or ultra-rapid metabolizer phenotype. All mITT participants with a completed PROMIS depression survey at 6 months are include. Participants with an incomplete PROMIS depression survey are excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Depression - Immediate PGx Testing (Modified Intent to Treat, mITT) | Depression - Delayed PGx Testing (Modified Intent to Treat, mITT)
Number analyzed (Participants) | 317 | 310
Participants | 153 | 122
Statistical Analysis 1: Comparison: Depression - Immediate PGx Testing (Modified Intent to Treat, mITT) vs Depression - Delayed PGx Testing (Modified Intent to Treat, mITT); Test type: Superiority; p = 0.0246, Chi-squared

6. Secondary Outcome: Number of Participants With Depression Remission as Measured by the Patient Health Questionnaire (PHQ-8)
Description: The PHQ-8 scores range from 0 to 24 and remission is defined as having a PHQ-8 score of ≤ 4.
Time Frame: 6 months
Population: Modified intent to treat (mITT) population consisting of participants with a CYP2C19 poor, rapid, or ultra-rapid metabolizer phenotype or a CYP2D6 poor or ultra-rapid metabolizer phenotype. All mITT participants with a completed PHQ-8 survey at 6 months are include. Participants with an incomplete PHQ-8 survey are excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Depression - Immediate PGx Testing (Modified Intent to Treat, mITT) | Depression - Delayed PGx Testing (Modified Intent to Treat, mITT)
Number analyzed (Participants) | 318 | 309
Participants | 95 | 65
Statistical Analysis 1: Comparison: Depression - Immediate PGx Testing (Modified Intent to Treat, mITT) vs Depression - Delayed PGx Testing (Modified Intent to Treat, mITT); Test type: Superiority; p = 0.0111, Chi-squared

7. Secondary Outcome: Number of Participants With 50% Reduction in Patient Health Questionnaire (PHQ-8) Score
Time Frame: 3 months
Population: Modified intent to treat (mITT) population consisting of participants with a CYP2C19 poor, rapid, or ultra-rapid metabolizer phenotype or a CYP2D6 poor or ultra-rapid metabolizer phenotype. All mITT participants with a completed PHQ-8 survey at baseline and 3 months are included. Participants with an incomplete PHQ-8 survey at either baseline or 3 months are excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Depression - Immediate PGx Testing (Modified Intent to Treat, mITT) | Depression - Delayed PGx Testing (Modified Intent to Treat, mITT)
Number analyzed (Participants) | 327 | 321
Participants | 92 | 71
Statistical Analysis 1: Comparison: Depression - Immediate PGx Testing (Modified Intent to Treat, mITT) vs Depression - Delayed PGx Testing (Modified Intent to Treat, mITT); Test type: Superiority; p = 0.0776, Chi-squared

8. Secondary Outcome: Number of Participants With Drug-gene Concordance
Description: Concordance defined as agreement between the PGx phenotype and SSRI medications reported.
Time Frame: 3 months
Population: Modified intent to treat (mITT) population consisting of participants with a CYP2C19 poor, rapid, or ultra-rapid metabolizer phenotype or a CYP2D6 poor or ultra-rapid metabolizer phenotype. All mITT participants with a completed medication review at 3 months are included. Participants without a medication review at 3 months are excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Depression - Immediate PGx Testing (Modified Intent to Treat, mITT) | Depression - Delayed PGx Testing (Modified Intent to Treat, mITT)
Number analyzed (Participants) | 323 | 315
Participants | 273 | 234
Statistical Analysis 1: Comparison: Depression - Immediate PGx Testing (Modified Intent to Treat, mITT) vs Depression - Delayed PGx Testing (Modified Intent to Treat, mITT); Test type: Superiority; p = 0.0014, Chi-squared

ADVERSE EVENTS:
Time Frame: Up to 6 months
Description: Per the study protocol, only Adverse Device Effect (ADE) events suspected to be related to the specimen collection, laboratory assay genotyping results, and phenoconversion recommendations from the Best Practice Alerts (BPAs)/Consult notes were reported to the IRB. Reportable ADEs or unanticipated Adverse Device Effect (UADEs) events including unanticipated study related deaths will be collected in the study database per IRB reporting policies. Medication side effects were not collected.
Arm/Group | Depression - Immediate PGx Testing | Depression - Delayed PGx Testing
All-Cause Mortality (participants affected / at risk) | 1/727 | 2/733
Serious Adverse Events (participants affected / at risk) | 0/727 | 0/733
Other Adverse Events (participants affected / at risk) | 0/727 | 0/733

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-05-23): https://cdn.clinicaltrials.gov/large-docs/55/NCT05966155/Prot_SAP_001.pdf
  • Informed Consent Form (2023-07-14): https://cdn.clinicaltrials.gov/large-docs/55/NCT05966155/ICF_000.pdf